CLINICAL TRIAL: NCT03081910
Title: Phase 1 Therapy With Manufactured Autologous T-Cells Expressing a Second Generation Chimeric Antigen Receptor (CAR) for Treatment of T-Cell Malignancies Expressing CD5 Antigen
Brief Title: Autologous T-Cells Expressing a Second Generation CAR for Treatment of T-Cell Malignancies Expressing CD5 Antigen
Acronym: MAGENTA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rayne Rouce, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-40466, MAGENTA; P50CA126752 (NIH)
Record Dates: First submitted 2017-03-08; First posted 2017-03-16 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: T-cell Acute Lymphoblastic Lymphoma; T-non-Hodgkin Lymphoma; T-cell Acute Lymphoblastic Leukemia
Keywords: Autologous CAR T cells; T-cell acute lymphoblastic lymphoma; T-non-Hodgkin Lymphoma; T-cell Acute Lymphoblastic Leukemia; Allogeneic CAR T cells
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autologous CD5.CAR/28zeta CAR T cells (Group A) - NOW CLOSED (Experimental): Three dose levels will be evaluated. The T cells will be administered with Cytoxan and fludarabine.If patients have experienced either a partial response or stable disease and completed the 6 week toxicity evaluation without evidence of DLT or other infectious complications, they will be eligible to receive up to 3 additional infusions of CD5 CAR.T cells. Patients remain eligible for up to 3 additional infusions as long as they continue to have a clinical response and absence of safety concerns. If patients experience a complete response following an additional infusion, investigators will recommend they proceed to allogeneic HSCT.
  Once dose escalation is completed, the trial will be expanded and treat up to an additional 6 patients (2 cohorts) at the MTD in each group to gather additional safety data and preliminary efficacy data.
  Interventions: Genetic: Autologous CD5.CAR/28zeta CAR T cells
- Allogeneic CD5.CAR/28zeta CAR T cells (Group B) (Experimental): Three dose levels will be evaluated. The T cells will be administered with Cytoxan and fludarabine.If patients have experienced either a partial response or stable disease and completed the 6 week toxicity evaluation without evidence of DLT or other infectious complications, they will be eligible to receive up to 3 additional infusions of CD5 CAR.T cells. Patients remain eligible for up to 3 additional infusions as long as they continue to have a clinical response and absence of safety concerns. If patients experience a complete response following an additional infusion, investigators will recommend they proceed to allogeneic HSCT.
  Once dose escalation is completed, the trial will be expanded and treat up to an additional 6 patients (2 cohorts) at the MTD in each group to gather additional safety data and preliminary efficacy data.
  Interventions: Genetic: Allogeneic CD5.CAR/28zeta CAR T cells

INTERVENTIONS:
Genetic: Autologous CD5.CAR/28zeta CAR T cells — Three dose levels will be evaluated:
  Dose level one: 1×10^7 cells/m2
  Dose level two: 5×10^7 cells/m2
  Dose level three: 1×10^8 cells/m2
  Arms: Autologous CD5.CAR/28zeta CAR T cells (Group A) - NOW CLOSED
Genetic: Allogeneic CD5.CAR/28zeta CAR T cells — Three dose levels will be evaluated:
  Dose level one: 1×10^7 cells/m2
  Dose level two: 5×10^7 cells/m2
  Dose level three: 1×10^8 cells/m2
  Arms: Allogeneic CD5.CAR/28zeta CAR T cells (Group B)

SUMMARY:
Patients eligible for this study have a type of blood cancer called T-cell leukemia or lymphoma (lymph gland cancer).

The body has different ways of fighting infection and disease. No one way seems perfect for fighting cancers. This research combines two different ways of fighting disease, antibodies and T cells. Antibodies are proteins that protect the body from bacterial and other diseases. T cells, or T lymphocytes, are special infection-fighting blood cells that can kill other cells including tumor cells. Both antibodies and T cells have shown promise treating patients with cancers, but have not been strong enough to cure most patients.

T lymphocytes can kill tumor cells but there normally are not enough of them. Some researchers have taken T cells from a person's blood, grown more in the lab then given them back to the person. In some patients who've had recent bone marrow or stem cell transplant, the number of T cells in their blood may not be enough to grow in the lab. In this case, T cells may be collected from their previous transplant donor, who has a similar tissue type.

The antibody used in this study, called anti-CD5, first came from mice that have developed immunity to human leukemia. This antibody sticks to T-cell leukemia or lymphoma cells because of a substance on the outside of these cells called CD5. CD5 antibodies have been used to treat people with T-cell leukemia and lymphoma. For this study, anti-CD5 has been changed so that instead of floating free in the blood it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor. In the lab, investigators have also found that T cells work better if stimulating proteins, such as one called CD28, are also added. Adding the CD28 makes the cells grow better and last longer in the body, giving them a better chance of killing the leukemia or lymphoma cells.

In this study investigators will attach the CD5 chimeric receptor with CD28 added to it to the patient's T cells or the previous bone marrow transplant donor's T cells. The investigators will then test how long the cells last. The decision to use the bone marrow transplant donor's T cells instead of the patient's will be based on 1) whether there is an available and willing donor and 2) the likelihood of the patient's T cells being able to grow in the lab. These CD5 chimeric receptor T cells with CD28 are investigational products not approved by the FDA.

UPDATE: Please note that the Autologous Arm of this study is now closed.

DETAILED DESCRIPTION:
To make the T cells the investigators will take blood from the patient or from the previous bone marrow transplant donor and stimulate it with growth factors to make the T cells grow. To get the CD5 antibody and CD28 to attach to the surface of the T cell, investigators insert the antibody gene into the T cell. This is done with a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell. This virus also helps investigators find the T cells in the patient's blood after they are injected. Because the patient will have received cells with a new gene in them the patient will be followed for a total of 15 years to see if there are any long term side effects of gene transfer.

When the patient is enrolled on this study, they will be assigned a dose of CD5 chimeric receptor-T cells Several studies suggest that the infused T cells need room to be able to proliferate (grow) and accomplish their functions and that this may not happen if there are too many other T cells in circulation. Because of that, the patient will receive two chemotherapy medications prior to receiving the CD5 chimeric receptor-T cells.

One medication is called cyclophosphamide and the other fludarabine. The patient will receive 3 daily doses of each drug, ending at least one day before the patient receives the chimeric receptor-T cells. These drugs will decrease the numbers of the patient's own T cells before the CD5 chimeric receptor T cells are infused and also will help decrease the number of other cells that may interfere with the chimeric receptor-T cells working well. These drugs are part of many regimens that are used to treat leukemia or lymphoma and not expected to have any effect on the patient's tumor with the doses given.

A potential side effect of receiving the chemotherapy as well as receiving CD5.CD28 Chimeric Receptor T cells is that it can cause development an Epstein Barr Virus (EBV) infection which can cause illness or formation of a growth or tumor. This side effect can be life threatening or fatal. To decrease this risk, following the chemotherapy but before administration of the CD5.CD28 Chimeric Receptor T cells, a dose of Rituximab (or a similar drug) will be given. Rituximab is an IV medication that is approved by the Food and Drug Administration to treat elevated levels of EBV in the body.

The patient will be given an injection of CD5.CD28 Chimeric Receptor T cells into the vein through an IV at the assigned dose. The injection will take from 1 to 10 minutes. Before the patient receives the injection, they may be given a dose of Benadryl and Tylenol. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

The patient will be followed in the clinic after the injection for up to 3 hours, and the patient will have to remain locally for a minimum of 6 weeks after the infusion. If there is evidence of EBV reactivation, the patient must remain locally for 8 weeks. During this initial phase patients will come to the clinic at least twice a week. Patients will be monitored closely for any side effects including signs of viral infection, or overgrowth of virus-infected cells that can behave like a tumor and require specific treatment. These side effects may require hospitalization for evaluation and management.

If after a 4-6 week evaluation period after the infusion, the patient has achieved a complete response (measured by bone marrow or radiology scans), the patient's primary oncology doctors may decide the patient should proceed to bone marrow transplant, at which time the patient will be removed from the treatment portion of the study.

Before being treated, the patient will receive a series of standard medical tests:

Physical exam and History; Blood tests to measure blood cells, kidney and liver function; Pregnancy test for female patients who are of child bearing potential; Measurements of the patient's tumor by scans and/or bone marrow studies

The patient will also receive standard medical tests during treatment and after:

Physical exams and History; Blood tests to measure blood cells, kidney and liver function; Blood tests to check for any evidence of viral infection

Graft versus Host Disease assessments:

Measurements of the patient's tumor by scans and/or bone marrow studies 6-8 weeks after the infusion and then per standard of care.

To learn more about the way the CD5 chimeric receptor-T cells are working and how long they last in the body, extra blood will be drawn. The total amount on any day is about 10 teaspoons (50 mL) or no more than 3 mL per 2.2 pounds body weight in children. This volume is considered safe but may be decreased if the patient is anemic. This blood may be drawn from a central line if the patient has one. Blood will be taken before the chemotherapy drugs, several hours after the T cell infusion, at 1 week, 2 weeks, 3 weeks (optional), 4 weeks, 6 weeks and 8 weeks (optional) after the infusion, at 3 months, 6 months, 9 months, at 1 year, every 6 months for 4 years, then yearly for a total of 15 years. We will also test blood to check for signs of viral infection at the following time points: within 1 to 2 weeks prior to chemotherapy drugs, prior to T cell infusion, then at weeks 1, 2, 3, 4, 6, 8 for all patients, and months 3, 6, 9, 12 for patients who do not proceed to bone marrow transplant. The total blood drawn during participation in this study will not exceed 280 teaspoons.

Once the dose escalation portion of the study is completed, the trial will be expanded and treat up to an additional 6 patients (2 cohorts) at the MTD in each group to gather additional safety data and preliminary efficacy data.

UPDATE: Please note that the Autologous Arm of this study is now closed.

ELIGIBILITY:
Procurement Inclusion Criteria for the Patient

Referred patients (Group A - NOW CLOSED) or their previous HSCT donors (Group B) will initially be consented for procurement of blood for generation of the transduced ATL. Patient eligibility criteria at this stage include:

1. Diagnosis of recurrent T-cell acute lymphoblastic leukemia (T-ALL), T-cell acute lymphoblastic lymphoma (T-LLy), or T-non-Hodgkin lymphoma (T-NHL, including Angioimmunoblastic T-cell lymphoma (AITL), Enteropathy-associated T-cell lymphoma (EATL), Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL), Peripheral T-cell lymphoma (PTCL) NOS, Anaplastic large cell lymphoma (ALCL), Adult T-cell leukemia/lymphoma, T cell prolymphocytic leukemia with symptomatic disease, Extranodal NK/T cell lymphoma, Mycosis fungoides/ Sezary Syndrome Stage IIB or higher))

   AND

   Group A (auto arm - NOW CLOSED): Transplant naïve or relapsed post-allogeneic HSCT OR

   Group B (allo arm): Relapsed post-allogeneic HSCT with previous HSCT donor from whom allogeneic MAGENTA CAR T cells can be manufactured

   AND
   * Suitable for allogeneic hematopoietic stem cell transplant (HSCT) with confirmation of an identified eligible allo-HSCT donor by FACT accredited institution
   * Confirmation that the center plans to proceed with transplant if CD5.CAR treatment induces a complete remission.

     * For T-NHL subjects, eligibility will be confined to disease stages where allogeneic HSCT is indicated.
2. CD5-positive tumor (result can be pending at this time). > 50% CD5 + blasts by flow cytometry or immunohistochemistry (tissue) assessed by a CLIA certified Flow Cytometry/Pathology laboratory.
3. Age ≤75 years old. NOTE: The first six (6) patients treated on the study should be adults (>18 yrs of age).
4. Life expectancy of greater than 12 weeks.
5. Patients must have an available partially-HLA matched allogeneic EBV-specific T cell line on a BCM IRB approved protocol which can be used as treatment in the event of uncontrolled EBV reactivation
6. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.
7. Hgb greather than or equal to 7.0 g/dL (can be transfused)
8. If pheresis required to collect blood:

   * Creatinine <1.5 × upper limit normal
   * AST <1.5 × upper limit normal
   * PT and APTT <1.5 × upper limit normal

Procurement Exclusion Criteria for the Patient (Group A)

1. Active infection requiring antibiotics.
2. Active infection with HIV
3. History of other cancer (except non-melanoma skin cancer or in situ breast cancer or cervix cancer) unless the tumor was successfully treated with curative intent at least 2 years before trial entry.

Procurement Inclusion Criteria for Normal Healthy Donor (Group B):

1. Donor must be prior hematopoietic stem cell transplant donor for patients relapsed post-allogeneic HSCT. Prior transplant donors will be screened with the standard blood bank donor questionnaire, medical history, and testing for infectious disease markers (IDMs; which may be pending at the time of blood collection). Medical history may be obtained by the patient's primary/referring transplant team if collection is being done remotely. The physician assessment, donor questionnaire, and IDMs will be reviewed by the principle investigator or appropriate designee to confirm/provide final eligibility determination and documented in the donor's medical record.
2. Informed consent explained to, understood by and signed by donor/LAR. Donor/LAR given copy of informed consent.

Treatment Inclusion Criteria

Patients must meet the following eligibility criteria to be included for treatment:

1. Diagnosis of recurrent T-cell acute lymphoblastic leukemia (T-ALL), T-cell acute lymphoblastic lymphoma (T-LLy), or T-non-Hodgkin lymphoma (T-NHL, including Angioimmunoblastic T-cell lymphoma (AITL), Enteropathy-associated T-cell lymphoma (EATL), Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL), Peripheral T-cell lymphoma (PTCL) NOS, Anaplastic large cell lymphoma (ALCL), Adult T-cell leukemia/lymphoma, T cell prolymphocytic leukemia with symptomatic disease, Extranodal NK/T cell lymphoma, Mycosis fungoides/ Sezary Syndrome Stage IIB or higher))

   AND

   Group A (auto arm - NOW CLOSED): Transplant naïve or relapsed post-allogeneic HSCT OR

   Group B (allo arm): Relapsed post-allogeneic HSCT with previous HSCT donor from whom allogeneic MAGENTA CAR T cells can be manufactured

   AND
   * Suitable for allogeneic hematopoietic stem cell transplant (HSCT) with confirmation of an identified eligible allo-HSCT donor by FACT accredited institution
   * Confirmation that the center plans to proceed with transplant if CD5.CAR treatment induces a complete remission.

     * For T-NHL subjects, eligibility will be confined to disease stages where allogeneic HSCT is indicated.
2. CD5-positive tumor. >50% CD5 + blasts by flow cytometry or immunohistochemistry (tissue) assessed by a CLIA certified Flow Cytometry/Pathology laboratory.
3. Age <75 years old. NOTE: The first six (6) patients treated on the study should be adults (>18 yrs of age).
4. Bilirubin less than 3 times the upper limit of normal.
5. AST less than 5 times the upper limit of normal.
6. Estimated GFR > 60 mL/min.
7. Pulse oximetry of > 90% on room air.
8. Karnofsky or Lansky score of ≥ 60%.
9. Recovered from acute toxic effects of prior chemotherapy at least one week before entering this study.
10. ≥ 60 days post-allogeneic HSCT at time of treatment.
11. Patients must have an available partially-HLA matched allogeneic EBV-specific T cell line on a BCM IRB approved protocol which can be used as treatment in the event of uncontrolled EBV reactivation.
12. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
13. Informed consent explained to, understood by, and signed by patient/guardian. Patient/guardian given copy of informed consent.

Treatment Exclusion Criteria

1. Currently receiving any investigational agents or having received any tumor vaccines within the previous 6 weeks.
2. History of hypersensitivity reactions to murine protein-containing products.
3. Pregnant or lactating.
4. Tumor in a location where enlargement could cause airway obstruction.
5. Active infection with HIV.
6. Clinically significant viral infection or uncontrolled viral reactivation of EBV, CMV, Adv, BK-virus, or HHV-6.
7. Evidence of acute GVHD > Grade II or active chronic GVHD > mild global severity score
8. Currently taking corticosteroids for therapy of GVHD at a dose of >0.5mg/kg prednisone equivalent
9. Patients who have received Immunosuppressive Treatment (IST) for GVHD within 28 days of infusion
10. Patients who have received donor lymphocyte infusion (DLI) within 28 days of infusion
11. Any of the following cardiac criteria: Atrial fibrillation/flutter; Myocardial infarction within the last 12 months; Prolonged QT syndrome or secondary prolonged QT, per investigator discretion. Cardiac echocardiography with LVSF<30% or LVEF<50%; or clinically significant pericardial effusion. Cardiac dysfunction NYHA III or IV (Confirmation of absence of these conditions within 12 months of treatment)
12. CNS abnormalities: Presence of CNS-3 disease defined as detectable cerebrospinal blast cells in a sample of CSF with ≥ 5 WBCs per mm3; History or presence of any CNS disorder such as a uncontrolled seizure disorder, cerebrovascular ischemia/hemorrhage within prior 6 months, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2040-09-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) rate | 6 weeks post-infusion
  Defined as the proportion of subjects in each group with DLT evaluated as per the CTCAE 4.0 with the exception of Cytokine Release Syndrome (CRS) and neurological toxicities that are related to T cell infusions.

SECONDARY OUTCOMES:
Overall Response Rate | 4 weeks pre-infusion and 6 weeks post-infusion
  Overall response rate is calculated as the proportion of subjects with the best overall response according to a revised response criteria for malignant lymphoma or bone marrow analyses for leukemia. Evaluations of tumor size will be performed within 4 weeks of beginning treatment and 6-8 weeks after T cell infusion (earlier if clinically indicated).

CONTACTS AND LOCATIONS:
Overall Officials: Rayne Rouce, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Dai Z, Mu W, Zhao Y, Jia X, Liu J, Wei Q, Tan T, Zhou J. The rational development of CD5-targeting biepitopic CARs with fully human heavy-chain-only antigen recognition domains. Mol Ther. 2021 Sep 1;29(9):2707-2722. doi: 10.1016/j.ymthe.2021.07.001. Epub 2021 Jul 16. PMID 34274536